CLINICAL TRIAL: NCT05408182
Title: Feasibility and Outcomes of an Early Discharge Protocol for Robotic Colorectal Surgery (eRCS): a Prospective Observational Study Open to International Collaboration
Brief Title: Early Discharge After Robotic Colorectal Surgery (eRCS): a Prospective Observational Study
Acronym: eRCS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ospedale di Camposampiero (Other)
Responsible Party: Principal Investigator, Stefan Morarasu, Principal Investigator, Ospedale di Camposampiero
Other Study IDs: OCamposampiero
Record Dates: First submitted 2022-05-26; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Colorectal Cancer; Surgery-Complications
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Perioperative Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Robotic colorectal resection with ERAS (or eRCS) perioperative care — All patients will undergo robotic colorectal resections using the Da Vinci xi system. All common colorectal procedures will be included: right/left colectomy, sigmoid colectomy, anterior resection with PME/TME/TaTME. Patient will undergo an enhanced recovery pathway perioperatively ensuring prompt recovery and early discharge. Most ERAS guidelines will be followed including preoperative nutrition, behavioral training, avoidance of drains, NG tubes, catheters, opioids, patient based volume repletion, wound local anesthetic infiltration, early mobilization, early postoperative feeding, spirometry and physiotherapy.

SUMMARY:
The enhanced recovery after surgery (ERAS) scheme has improved recovery of patients by addressing the surgical stress and enabling a proactive perioperative care which has proven to decrease postoperative complications and reduce hospital stay. ERAS had a major beneficial effect in open colorectal surgery, while in laparoscopic surgery the additional benefit was somewhat less. Also, current literature is not clear if ERAS can improve operative outcomes of robotic colorectal surgery.

Starting from the already proven ERAS protocol, we aim to build a selective enhanced recovery scheme and a standardized early follow-up pathway enabling early safe discharge of low-risk patients after robotic colorectal surgery. This observational study will also design and assess the feasibility and clinical outcomes of an Early discharge Colorectal Surgery (eRCS) protocol which may be used to discharge patients in postoperative day 1 after robotic colorectal resections through close virtual and outpatient follow-up.

DETAILED DESCRIPTION:
This is a prospective observational study open to collaboration with international centers with expertise in robotic colorectal surgery. The cohort will include adult patients, categorized as low risk based on the inclusion criteria, which will undergo elective colorectal surgery under the governance of ERAS to enable early discharge. Patient will be followed-up clinically through pain scores, mobility scores, satisfaction and postoperative outcomes (e.g., surgical site infections, leaks, ileus, readmissions) to assess their recovery within the first 30 days postoperatively. The subgroup of patients which will be discharged on postoperative day 1 (POD 1) will form the 24h surgery group. These patients will also be closely followed-up virtually and through the outpatient department for blood samples and clinical examination.

All data on patients including follow-up data will be recorded in an encrypted Excel database. Patient will be followed-up according to the above plan up to 30 days postoperatively, when they will be asked to fill in a questionnaire to assess patient reported experience (VAS score, mobility score and satisfaction rate). Postoperative complications and readmissions will be recorded.

Main outcomes:

* Postoperative day of discharge (early 1, intermediate 2, standard 3-5)
* Patient reported outcomes: pain score (VAS), mobility score, nausea score, food tolerance score, satisfaction rate during admission, on day of discharge, on days 2, 4 and 7 for patient discharged on POD 1 and for all patients at POD 30
* Postoperative complications: surgical site infection, urinary infection, other source of sepsis, ileus, intraabdominal sepsis, anastomotic leak, cardiovascular complications, respiratory complications
* Readmission rate, reintervention rate

ELIGIBILITY:
Inclusion Criteria:

* Age less than 75yo
* ASA grade I and II
* Not on anticoagulation
* Elective colorectal resections
* Does not require stoma
* No intraoperative complications (surgical team happy with procedure)
* Patient/Caregiver thoroughly counselled about the aim and each step of the protocol (for patients which will be discharged on POD 1)
* Patient/Caregiver understands what to expect and knows how to manage possible issues (for patients which will be discharged on POD 1)
* Patient/Caregiver has a direct line to the Nurse Practitioner/Surgical team member (for patients which will be discharged on POD 1)
* Able to attend virtual and clinic follow-up in the first 10 days postoperatively (transport to hospital available - for patients which will be discharged on POD 1)

Exclusion Criteria:

* Age more than 75yo
* ASA grade III
* Patient on anticoagulation
* Emergency surgery
* Requires stoma
* Intraoperative complications: iatrogenic injuries, significant bleeding, anaesthetic issues, new significant pathology encountered, complicated procedure, conversion to open surgery
* Patient/Caregiver refuses early discharge
* Caregiver not available to support patient at home (for patients which will be discharged on POD 1)
* Cannot attend virtual or/and clinical follow-up if discharged on POD 1

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The cohort will include adult patients, categorized as low risk based on the inclusion criteria which will undergo elective colorectal surgery under the governance of ERAS to enable early discharge.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Days of hospitalization | 30 days
  The length of stay in hospital will be recorded in number of days
Postoperative pain score | 30 days
  Level of postoperative pain will be recorded through the Visual Assessment Scale (VAS). Patient will score level of pain from 1 (no pain) to 10 (worst pain ever felt). Pain will be recorded on postoperative days 1, 2, 3, 5, 7 and 30. Pain score will be measured at rest and when patient is mobilizing.

SECONDARY OUTCOMES:
Mobility score | 30 days
  Level of mobility will be recorded at postoperative days 1, 2, 3 and day of discharge (if > 72h). Mobility scale: 0 = not mobilizing; 1 = able to walk with assistance; 2 = able to walk without assistance; 3 = caring for himself with assistance; 4 = caring for himself independently; 5 = fully independent, but not as before the operation; 6 = fully independent, similar to before the operation
Post discharge satisfaction | 30 days
  Patient reported satisfaction with treatment will be measured on the 3rd day after discharge (if patient was discharged before postoperative day 3) and/or at 30 days postoperatively.
  Satisfaction scale at initial post discharge assessment: 1 = unhappy with current plan/requests readmission; 2 = feels should have stayed longer in hospital, but will manage at home; 4 = now he is happy with plan/early discharge, but initially unhappy; 5 = happy with plan/early discharge
  Satisfaction scale at 30 days postoperatively: 1 = unhappy with care; 2 = unhappy, feels should have stayed longer in hospital; 4 = unhappy, feels should have been more closely followed-up; 5 = initially was unhappy, but now feels management plan was appropriate; 6 = happy with care received
Overall Morbidity | 30 days
  Overall morbidity will be recorded considering surgical complications (surgical site infection, anastomotic leak, abdominal sepsis, ileus, postoperative bowel obstruction, bleeding)
Readmission rate | 30 days
  Readmissions in the first 30 days postoperatively will be recorded. Duration of inpatient stay during readmission and type of management (e.g., reintervention, invasive procedure such as interventional radiology, medical care) will be described.

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Morpurgo, Principal Investigator — Department of Surgery Hospital Camposampiero Azienda ULSS 6 Euganea
Locations (1):
- Camposampiero Hospital, Camposampiero, Padova, Italy

IPD SHARING:
Plan to Share IPD: Undecided